CLINICAL TRIAL: NCT04953585
Title: Effectiveness of Managing Suspected Metastasis and Progress Using Plasma D-dimer Testing in Gastric Cancer Patients
Acronym: EMPUPDTGCP
Status: Completed | Type: Observational
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Other Study IDs: NO.81501826
Record Dates: First submitted 2021-06-15; First posted 2021-07-08 (Actual); Last update posted 2021-07-08 (Actual); Status verified 2021-01

CONDITIONS: Stomach Neoplasms
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — the pathological specimen after surgical resection
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Normal D-dimer group: preoperative plasma D-dimer levels less than or equal to 1mg/L
  Interventions: Procedure: radical gastrectomy
- Elevated D-dimer group: preoperative plasma D-dimer levels greater than 1mg/L
  Interventions: Procedure: radical gastrectomy

INTERVENTIONS:
Procedure: radical gastrectomy — According to the size and location of the tumor, the appropriate surgical method was selected for radical gastrectomy

SUMMARY:
For prognosis evaluation, investigators enroll gastric cancer patients who underwent radical gastrectomy and collect the laboratory examination and clinicopathological characteristics. Then independent risk factors for overall survival will be analysed. For predicting efficacy evaluation, investigators also collect information of patients first diagnosed with metastases. Diagnostic efficacy is analysed by receiver operator characteristic curve method.

DETAILED DESCRIPTION:
To investigate the novel predictive value of coagulation factors for postoperative outcomes after radical gastrectomy in patients with gastric cancer, investigators enroll patients with a pathologically confirmed diagnosis of gastric cancer who underwent radical gastrectomy between January 2021 and february 2017. Patients follow up data were obtained by regular follow-up. The most recent preoperative laboratory tests and clinicopathological characteristics were evaluated. Patients are devided into two groups according to our target indicator. The 5-year overall survival rate is analysed by Kaplan-Meier method. The independent risk factors for overall survival are analysed by Cox proportional hazard regression method. Investigators hypothesized that the target factor is closely related to disease progression. Whether it can be used as a tumor marker to predict metastasis is to be studied. Investigators collect laboratory examination including tumor markers of patients first diagnosed with metastases. Diagnostic efficacy is analysed and compared by receiver operator characteristic curve method.

ELIGIBILITY:
Inclusion Criteria:

* all patients were newly diagnosed with gastric cancer;
* all patients were pathologically diagnosed;
* all patients had pre-treatment coagulation test;
* stage I-IV disease;
* age≥18 years

Exclusion Criteria:

* accompanying or secondary to other tumors;
* had history of venous thrombosis or received any anti-coagulation treatment;
* acute infection or intravascular disseminated coagulation;
* pregnancy or lactation;
* history of neoadjuvant chemotherapy;
* Lost to follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients first diagnosed with gastric cancer and suitable for radical resection
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
overall survival time | From date of radical gastrectomy until the date of last follow-up or date of death from gastric cancer, whichever came first, assessed up to 48 months
  From date of radical gastrectomy until the date of last follow-up or date of death from gastric cancer, whichever came first, assessed up to 48 months

CONTACTS AND LOCATIONS:
Overall Officials: Dongmei Diao, Study Chair — First Affiliated Hospital Xi'an Jiaotong University
Locations (1):
- The First Affiliated Hospital of Xi 'an Jiaotong University, Xi'an, Shaanxi, China